CLINICAL TRIAL: NCT03263741
Title: Exploratory Study on the Efficiency and Safety of Paclitaxel + S-1 + Oxaliplatin Chemotherapy in the Patients With Locally Advanced or Advanced Gastric Cancer
Brief Title: Exploratory Study on the Paclitaxel + S-1 + Oxaliplatin (PSOX) for Locally Advanced or Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Qinghai University (Other)
Responsible Party: Principal Investigator, Jiuda Zhao, Professor, Affiliated Hospital of Qinghai University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHQU-2017002
Record Dates: First submitted 2017-08-22; First posted 2017-08-28 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Gastric Cancer
Keywords: Paclitaxel; S-1; Oxaliplatin; Efficiency; safety
MeSH Terms: conditions — Stomach Neoplasms | interventions — Paclitaxel; S 1 (combination); Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Paclitaxel + S-1 + Oxaliplatin group (Experimental): Paclitaxel: 135 mg/m2, iv, 3h, at D1 ; S-1: 40mg twice daily for patients with a body surface area (BSA) < 1.25 m2, 50mg twice daily for patients with a BSA of 1.25 m2 to < 1.5 m2, 60mg twice daily for patients with a BSA of ≥ 1.5 m2 for two weeks, and then suspend for one week; Oxaliplatin: 85 mg/m2, iv, 2h, at D1.
  Interventions: Drug: Paclitaxel + S-1 + Oxaliplatin

INTERVENTIONS:
Drug: Paclitaxel + S-1 + Oxaliplatin — Paclitaxel: 135 mg/m2, iv, 3h, at D1. S-1: S-1: 40mg twice daily for patients with a body surface area (BSA) < 1.25 m2, 50mg twice daily for patients with a BSA of 1.25 m2 to < 1.5 m2, 60mg twice daily for patients with a BSA of ≥ 1.5 m2 for two weeks, and then suspend for one week.
  Oxaliplatin: 85 mg/m2, iv, 2h, at D1.
  Other Names: Paclitaxel + S-1 + Oxaliplatin chemotherapy

SUMMARY:
Explore the Efficiency and Safety of Paclitaxel + S-1 + Oxaliplatin (PSOX) Chemotherapy in the Patients with Locally Advanced or Advanced Gastric Cancer

DETAILED DESCRIPTION:
To assess the Efficiency and safety of Paclitaxel + S-1 + Oxaliplatin(PSOX) in the Patients with Locally Advanced or Advanced Gastric Cancer

ELIGIBILITY:
Inclusion Criteria:

1. Histopathology or cytopathology proven gastric cancer or gastroesophageal adenocarcinoma;
2. Locally advanced, or recurrent, or metastasis disease；
3. Chemotherapy-naive or disease progress at least 6 months after adjuvant chemotherapy completed;
4. Life expectancy of at least 3 months;
5. ECOG score 0-1;
6. Age: 18~70 years old;
7. Normal hemodynamic indices before the recruitment (including blood cell count and liver/kidney function). For example: WBC>4.0×109/L, NEU >1.5×109/L, PLT>100×109/L, BIL<1.5 times of upper limit of normal reference value, ALT and AST<2.5 times of upper limit of normal reference value, and CRE<1.2mg/dl;
8. Good cardiac function before the recruitment, no seizure of myocardial infarction in past half year, and controllable hypertension and other coronary heart diseases;
9. Not concomitant with other uncontrollable benign diseases before the recruitment (e.g. the infection in the lung, kidney and liver);
10. Not participating in other study projects before and during the treatment;
11. Voluntarily signed the informed consent.

Exclusion Criteria:

1. Previously treated with first-line chemotherapy;
2. Allergy to the drugs in this protocol;
3. Pregnant or lactating women;
4. Women at childbearing age and of pregnancy desire during the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | 2 years
  The sum of complete remission (CR) rate and partial remission (PR) rate.

SECONDARY OUTCOMES:
Progression-free survival(PFS) | 2 years
  From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
Overall survival(OS) | 2 years
  From date of enrollment until the date of death from any cause, assessed up to 60 months
Disease control rate(DCR) | 2 years
  The sum of CR rate, PR rate and stable disease(SD) rate. Response will be measured through first-line treatment completion, up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jiuda Zhao, M.D., Principal Investigator — Affiliated Hospital of Qinghai University
Locations (1):
- Affiliated Hospital of Qinghai University, Xining, Qinghai, China